CLINICAL TRIAL: NCT03971058
Title: Characterisation of Cellular and Humoral Immune Responses Following the First Booster Immunisation With the Inactivated, Purified Japanese Encephalitis Vaccine IXIARO® in Elderly Compared to Young Individuals.
Brief Title: Immune Responses After a Booster Immunisation With IXIARO® in Elderly Compared to Young Individuals.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Valneva Austria GmbH (Industry)
Responsible Party: Principal Investigator, Univ. Prof. Dr. Ursula Wiedermann, Univ.-Prof. MD PhD, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IXIARO-booster senescence; 2016-002894-36 (EudraCT Number)
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Japanese Encephalitis Vaccine
Keywords: Japanese Encephalitis vaccine; immune responses

STUDY DESIGN:
Intervention Model Description: Immune Responses After a Booster Immunisation With IXIARO® in Elderly Compared to Young Individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- young individuals (Active Comparator): Immune Responses After a Booster Immunisation With IXIARO®- Japanese Encephalitis vaccine
  Interventions: Biological: IXIARO®- Japanese Encephalitis vaccine
- elderly individuals (Active Comparator): Immune Responses After a Booster Immunisation With IXIARO®- Japanese Encephalitis vaccine
  Interventions: Biological: IXIARO®- Japanese Encephalitis vaccine

INTERVENTIONS:
Biological: IXIARO®- Japanese Encephalitis vaccine — Booster Immunisation With IXIARO®- Japanese Encephalitis vaccine

SUMMARY:
The aim of this study is to investigate the immune responses following a booster immunisation with the Japanese Encephalitis vaccine in elderly subjects (above 60 years of age) in comparison to a young study group.

DETAILED DESCRIPTION:
The condition under investigation is the naturally aging immune system. The aim of this study is to investigate the immune responses following a booster immunisation with the Japanese Encephalitis vaccine in elderly subjects (above 60 years of age) in comparison to a young study group.Testing the difference of the JEV-antibody titre increase between young and elderly adults between visit 1 (before booster vaccination) and up to visit 4 (6 months after booster vaccination).

Testing cellular immunity (cytokine production after JEV as well as TBE stimulation) on visit 1, 2 (one week after booster immunisation) and 3 between both age groups.

Testing of surface markers of different T and B cell subsets before and after JE-booster vaccination (on visit 1-3) in comparison between both age groups.

Testing TBE-antibody titres before and after JE-booster vaccination (on visit 1-4) in both age groups.

Testing CMV serology at visit 1 in both age groups.

ELIGIBILITY:
Inclusion Criteria:

* participation in the preceeding study "IXIARO®-senescence" (EudraCTno: 2010-018630-52) without protocoll violation OR 2 documented IXIARO® vaccinations 28 days (-8/+ 30 days) apart between January 2010 and April 2014 at the age of 18 to 40 years or above the age of 60.
* good state of health including individuals with medically controlled minor underlying disease (such as hypertension, hypercholesterinemia, NIDDM)
* willingness to sign written informed consent

major Exclusion Criteria:

* Already received an booster (3rd dose) of IXIARO ®
* Vaccination with other JE vaccine (e.g. Je-vax)
* clinically manifest infection with another Flavivirus within 1 year prior study inclusion (yellow fever, Dengue fever, West Nile, TBE)
* past infection with the JEV
* vaccination against yellow fever, Dengue, West Nile within 6 months prior to study inclusion
* TBE vaccination within the last 30 days prior to study inclusion
* immunosuppressive therapy (intake>14d) within 30 days before IXIARO booster till V3 (day 42+/-4), Corticosteroids like Prednisolon > and = 20mg/day; allowed: topic or inhalative application
* immunodeficiency or st. p. organ transplantation
* autoimmune disease except vitiligo or diseases of the thyroid gland with thyroid hormon substitution therapy
* immuntherapy within 2 weeks before or after Ixiaro Booster
* current acute infection or exacerbation of a chronic illness
* cancer within the last 5 years
* clinically significant haematological, renal, pulmonary, hepatic, neurological, cardiovascular disease which is not treated adequately within 12 weeks before Ixiaro booster
* known infection with HIV, Hep B and Hep C
* Guillain - Barré- Syndrome (GBS) - anamnestic
* anamnestic anaphylaxie, atopy oder severe hypersensivity against ingredients of IXIARO
* drug abuse/alcohol abuse
* pregnancy and breastfeeding
* plasma donation within the last 4 months
* receiving blood or immunglobulins within 3 months before v1
* significant mental disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
JEV antibody titer increase/course between visit 1 (before the booster vaccination) and Visit 3 | Visit 3 day 42+/-4
  Testing the difference of the JEV antibodies increase between young and elderly adults between Visit 1 (before booster vaccination) and Visit 3 (day 42+/-4 after Booster vaccination)

SECONDARY OUTCOMES:
Testing the difference of the JEV antibody titer between young and elderly adults | Visit 1, day 0) till Visit 4 (day 168 +/- 14)
  Testing the difference of the JEV antibody titer before the booster vaccination with IXIARO® (Visite 1, day 0) till Visit 4 (day 168 +/- 14) in comparison between the age groups
Testing cellular immunity | Visit 1, day 0), seven days after booster vaccination (Visit 2, day 7 (+2).
  Testing cellular immunity (cytokine production of IL-2, IFN-g, TNF-alpha, IL-6, IL-10, IL-21 after stimulation with JEV antigen) before the booster vaccination with IXIARO® (Visit 1, day 0), seven days (Visit 2, day 7 (+2) after and after 42 days (Visit 3, day 42 (+/-4)) after that in comparison between the age groups.
Testing of lymphocyte populations with FACS analysis | Visit 1, day 0), seven days after booster vaccination (Visit 2, day 7 (+2) and 42 days (Visit 3, day 42 (+/-4) after booster vaccination
  Testing of lymphocyte populations via testing surface markers of different B and T cell subsets with FACS and bloodcount
Testing of CMV serology | Visit 1, day 0
  Testing of CMV Seropositivity at the time of the booster vaccination with IXIARO® at Visit 1 (day 0) in both age groups
TBE titer increase/course | Visit 1, day 0), seven days (Visit 2, day 7 (+2), 42 days (Visit 3, day 42 (+/-4) und 6 Months (Visit 4, day 168 (+/- 14)
  Tick borne encephalitis titer before booster vaccination with IXIARO® (Visit 1, day 0), seven days after the booster vaccination (Visit 2, day 7 (+2),and 42 days (Visit 3, day 42 (+/-4) after the booster vaccination and 6 months (Visit 4, day 168 (+/- 14) after the booster vaccination and the in comparison between age groups.
Testing of cellular immunity-Testing of cytokine production | Visit 1, day 0; Visit 2, day 7 (+2)
  Testing of cellular immunity (cytokine production of IL-2, TNF-alpha, IL-6, IL-10 after stimulation mit TBE Antigen) before and seven days after the booster vaccination with IXIARO® (Visit 1, day 0; Visit 2, day 7 (+2) in comparison between the age groups

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wiedermann-Schmidt, Univ Prof MD, Principal Investigator — Medical University of Vienna, ISPTM
Locations (2):
- Austria (2):
  - Medical University of Vienna, Vienna
  - Medical University Vienna, Institute of Specific Prophylaxis and Tropical Medicine, Vienna